CLINICAL TRIAL: NCT06930196
Title: Pain: A Century's Old Approach to Treatment With Objective Documentation
Brief Title: By Potentially Adding a Century Old Therapeutic Measure to Pain Treatment Regimens Called Osteopathic Manipulative Treatment, Can Help Decrease Muscle and Bone Pain and the Usage of Opioid Pain Medication.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Skagit Regional Health (Other)
Collaborators: Philadelphia College of Osteopathic Medicine (Other); University of Eastern Finland (Other)
Responsible Party: Principal Investigator, Precious L Barnes DO, MS, MS, Hospitalist Physician, Principal Investigator Board certified in Family medicine and Neuromusculoskeletal Medicine, Skagit Regional Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SkagitRegional
Record Dates: First submitted 2025-03-18; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Osteopathic Manipulative Treatment
Keywords: OMT; Osteopathic Manipulative Treatment; Non opioid pain management; Alternative pain management; Musculoskeletal medicine
MeSH Terms: interventions — Tocopherols

STUDY DESIGN:
Intervention Model Description: 3 arm model but the goal was 5
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The person who provided treatment and the person who operated the machine were blinded to each other. Participants did not know which treatment they were going to receive until it was actually performed. The Statistician used only deidentified data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Muscle Energy Treatment (Active Comparator): Subjects received Muscle Energy osteopathic manipulative treatment after analysis with the SA201 for somatic dysfunction and then again after treatment.
  Interventions: Other: Muscle Energy; Device: The Ultralign SA201 used for measuring tissue texture changes; Device: IsoTouch
- High Velocity Low Amplitude (Active Comparator): Subjects received High Velocity High Amplitude osteopathic manipulative treatment after analysis with the SA201 for somatic dysfunction and then again after treatment.
  Interventions: Other: High Velocity Low Amplitude; Device: The Ultralign SA201 used for measuring tissue texture changes; Device: IsoTouch
- Counterstrain (Active Comparator): Subjects received Counterstrain osteopathic manipulative treatment after analysis with the SA201 for somatic dysfunction and then again after treatment.
  Interventions: Other: Counterstrain; Device: The Ultralign SA201 used for measuring tissue texture changes; Device: IsoTouch

INTERVENTIONS:
Other: Counterstrain — Subjects were first analyzed for tissue texture changes with the SA201 then given an osteopathic treatment and analyzed post treatment with the SA201 to analyze for tissue texture changes.
  Other Names: Intervention number 3
  Arms: Counterstrain
Other: Muscle Energy — Subjects were first analyzed with the Ultralign SA201/Spineliner, then treated with an osteopathic technique, and then reassessed with the SA201 for tissue texture changes.
  Other Names: Intervention number 2
  Arms: Muscle Energy Treatment
Other: High Velocity Low Amplitude — Subjects were first analyzed for tissue texture changes with the SA201 then given an osteopathic treatment and analyzed post treatment with the SA201 to analyze for tissue texture changes.
  Other Names: Intervention number 1
  Arms: High Velocity Low Amplitude
Device: The Ultralign SA201 used for measuring tissue texture changes — The Ultralign SA201 was used for diagnostic purposes to measure the tissue texture changes of the paraspinal cervical muscles pre and post treatment
  Other Names: Ultraslign SA201; Spineliner; SA201
Device: IsoTouch — The IsoTouch is a palpation monitoring system that uses capacitance pressure sensors in the pads of gloves to measure the palpation pressures used for both diagnosis and treatment using OMT. No sensation is felt by either the subject or operator other than a feeling of a glove being used during treatment. No electrical impulses are sent or should be experienced by either party as the sensors are merely pads that sense pressure.
  Other Names: Palpation monitors

SUMMARY:
Osteopathic Manipulative Treatment (OMT) has been used to successfully treat patients for over a hundred years. Even though there have been many subjective clinical results, there is still little research measuring the actual mechanical change to a spinal segment produced by OMT or the actual palpatory changes that one is able to detect or elicit.

The Ultralign SA201System (also called a Spineliner internationally) is an advanced technical instrument commercially used for spinal analysis and treatment. It was originally designed to assist chiropractors in locating and correcting "subluxations" or "fixations", which may share many characteristics in common with "somatic dysfunction" or perhaps be identical in all but name. This system can analyze selected regions of the spine for comparison to adjacent tissues as well as pre and post treatment changes using computer graphics and actual digital numbers to describe the changes around a spinal segment. In this study, only the analysis part of the SA201 will be used.

The analytical function of the SA201 allows the user to place a force transducer (small, smooth, rubber-like rod) against the skin overlaying a subject's spine and release an impulse (gentle tap) into the somatic tissues of the underlying spinal segment. The force impulse is transmitted through the sensor to the underlying area, soft tissues and articular elements of the subject which results in the formation of a waveform that is characteristic of the ratio of tissue resistance and force dissipation. Interpretation of the waveform measured by the SA201's force sensor provides an indication of the "stiffness" or "compliance" of each spinal segment as well as its "hysteresis" (the lagging of an effect behind its cause or how quickly the tissues tested return towards their original condition). The shape of the wave may be analyzed and further interpreted to reflect muscle spasm or other underlying tissue conditions.

In this research study the investigators will obtain hysteresis measurements before and after treatment of spinal areas diagnosed by palpation to contain somatic dysfunction (SD). Hysteresis is the time it takes for the tissues to recoil after a deforming force has been introduced. Measurements of hysteresis will be taken using the SA201 before and after use of two OMT techniques used to relieve SD, High Velocity Low Amplitude (HVLA), Muscle Energy (ME) and Counterstrain (CS). Selection of these three techniques shall be randomized. The investigators will note if the SA201 is able to detect a difference in the hysteresis characteristics of a given SD and document whether OMT is capable of changing this objective parameter related to tissue texture; furthermore, a difference (if there is one) may be detected and quantified to determine if there is a different outcome between the different treatment modalities.

The investigators also used a pressure sensor system called the IsoTOUCH during the diagnosis/treatment in the study to gain a better understanding of the amount of pressure that the SA201uses to diagnose a SD compared to the diagnostic pressure the Palpator uses. The IsoTouch were a pair of gloves worn by the physician administering OMT. No sensation other than palpation with gloved fingers were felt by the patient.

At preset pressures, the SA201will document hysteresis characteristics of segments considered to have somatic dysfunction or not. This permits comparison of the dysfunctional, normal and corrected sites diagnosed by hand and the sites independently determined by the technology. It should also be able to graphically illustrate the change in the dysfunctional segment's response to the SA201 stimulus pre and post treatment, as well as to document if there is a difference between the various OMT treatment modalities. This machine also allows for the testing of more than one element simultaneously without compromising other aspects of the study.

While the SA201 and the IsoTouch palpation monitors are able to diagnosis all segments of the spine this study will limit diagnosis and treatment to the cervical spine only at this time. Later studies can potentially expand to the other areas of the spine and body.

DETAILED DESCRIPTION:
Subjects will randomly choose a number 1-3. The number correlates to one of three treatment techniques ME, CS, or HVLA. Prior to treatment subjects will be analyzed with the Ultralign SA201 to the cervical region only to assess the hysteresis of the segment. The subject will then go to another room and be treated with the OMT technique chosen prior to the start of the study. Post treatment the subject will then return to be reassessed by the Ultralign SA201 for post treatment analysis.

The Ultralign SA201 is able to measure tissue texture hysteresis using durometers. A durometer is a standardized way of measuring the hardness of materials like rubber or plastic. It is a measure of how resistant a plastic is to deformation caused by mechanical indentation or abrasion. Durometer measurement scales range from 0 to 100. This scale is commonly used to measure the plasticity of airplane wings to ensure that a plane is still in acceptable flight conditions. In this study we are looking at the changes in hysteresis of the cervical region (measured in durometers) to see if objective changes in the cervical region post OMT can be observed.

The physician treating the subjects and the physician operating the SA201 will remained blind to the others findings until the completion of the study. There by making this a partially blinded study. The Ultralign SA201 operator will also remain blind to the OMT technique used until completion of the study. By using the Ultralign SA201 it was projected that it would be able to detect tissue texture (hysteresis) changes objectively supporting the usage of OMT as an adjunctive treatment for treating pain.

Subjects will also do a pre and post treatment questionnaire using the Numeric Pain Rating scale to describe their pain (if any) along with noting their experience while being analyzed by the SA201. A 0 is no pain and a 10 is the worst pain.

Ultimately the pre and post treatment pain scales will be compared to see if there is a decrease in overall pain as well as to see if there is an overall change in hysteresis measurements (in durometers) in conjunction with the decrease in pain.

ELIGIBILITY:
Inclusion Criteria:

The subjects that will be sought for this study will be male or female subjects from the ages of 18-65 years. Because this is a one session study, where a person lives does not preclude them from participating in this study.

Healthy Volunteers are the volunteers that may present with or without a cervical somatic dysfunction, having a cervical somatic dysfunction is a common biomechanical occurrence and does not constitute a person as being unhealthy.

Exclusion Criteria:

1. Subjects younger than age 18 or over the age of 65 years.
2. History of abnormal findings on brain or cervical CT/MRI
3. History of diagnosis of symptomatic osteoarthritis of the cervical spine (as documented in previous imaging studies) or as evidenced by palpation and provocative tests during structural exam
4. Significant scoliosis that contributes to back or neck pain diagnosed by structural exam
5. Current diagnosis or history of depression, except for mild situational depression specifically diagnosed as associated with chronic headaches
6. Significant psychiatric disorders present or past including, but not limited to: borderline personality, bipolar disorder or schizophrenia
7. History of systemic disease which includes, but is not limited to: rheumatoid arthritis, Marfan's syndrome, fibromyalgia, Ehler-Danlos Syndrome or other connective tissue disease, lupus or ankylosing spondylitis
8. History of neoplastic disease
9. Involvement in current litigation involving the neuromusculoskeletal syndrome

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2011-06-01 (Actual); Primary Completion 2012-06-30 (Actual); Study Completion 2012-06-30 (Actual)

PRIMARY OUTCOMES:
Can tissue texture changes be objectively documented post OMT | 2 weeks
  Each subject will have paraspinal cerivcal musculoskeletal hysteresis measurements taken of the cervical spine (OA-C7) using the Ultralign SA201. The Ultralign SA201 measures tissue texture changes in durometers. The durometer readings will be compared pre and post osteopathic manipulative to see if the overall change in the somatic dysfunction. Changes in the durometer shows changes in the tissue.
  After the final collection of data an ANOVA data analysis of the durometer readings will be performed to see if there is an objective change in tissue hysteresis after osteopathic manipulative treatment has been administered.

SECONDARY OUTCOMES:
How much pressure is actually used during diagnosis and treatment | 2 weeks
  Palpation monitors will be used during diagnosis and treatment to observe the level of pressure used in pounds to assess reproducibility and consistency of each treatment and diagnosis. The palpation monitors will only be used during the diagnosis and treatment phase of OMT. The monitoring of this will allow for reproducibility and consistency to be shown with osteopathic manipulative treatment.
  The amount of pressure in pounds will be measured during both diagnosis and treatment to see the amount of diagnostic pressure used to diagnosis and treat a segment. By understanding this, it allows for better information for others who would like to reproduce this study but also for those in clinical practice to know how much or how little pressure is used during diagnosis and treatment. If activating forces show a very low pressure being used, then some treatments with low activating pressures may be able to be used in more delicate populations such as those with rheumatoid arthritis.

OTHER OUTCOMES:
Pain rating | Immediately before and after treatment
  A Pre and post treatment Numeric Rating Pain Scale questionnaire will be taken to assess cervical pain level as well as any discomfort that may have been caused by the Ultralign SA201. The main purpose of the questionnaire is to see if there is decreased reported neck pain post treatment in conjunction to objective cervical hysteresis changes.

CONTACTS AND LOCATIONS:
Locations (1):
- Philadelphia College of Osteopathic Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be shared
Supporting Information: Study Protocol, CSR
Time Frame: Starting 6 months after publication information will be shared
Access Criteria: Data information will be available to specified statisticians for ANOVA data analysis along with the investigators.

REFERENCES:
- [Background] Rehman Y, Ferguson H, Bozek A, Blair J, Allison A, Johnston R. Osteopathic Manual Treatment for Pain Severity, Functional Improvement, and Return to Work in Patients With Chronic Pain. J Am Osteopath Assoc. 2020 Dec 1;120(12):888-906. doi: 10.7556/jaoa.2020.128. PMID 32946545
- [Background] Jerome JA. An Osteopathic Approach to Chronic Pain Management. J Am Osteopath Assoc. 2017 May 1;117(5):306-314. doi: 10.7556/jaoa.2017.056. PMID 28459476
- [Background] Seffinger M. Foundations of Osteopathic Medicine. Fourth Edition. Wolters Kluwer; 2018.
- [Background] Licciardone JC, Schultz MJ, Amen B. Osteopathic Manipulation in the Management of Chronic Pain: Current Perspectives. J Pain Res. 2020 Jul 20;13:1839-1847. doi: 10.2147/JPR.S183170. eCollection 2020. PMID 32765058
- [Background] Barnes PL, Laboy F 3rd, Noto-Bell L, Ferencz V, Nelson J, Kuchera ML. A comparative study of cervical hysteresis characteristics after various osteopathic manipulative treatment (OMT) modalities. J Bodyw Mov Ther. 2013 Jan;17(1):89-94. doi: 10.1016/j.jbmt.2012.10.004. Epub 2012 Dec 5. PMID 23294689
- [Background] Kim G, St. Laurent E, Keane J, Goldstein L. Muscle dysfunction in head and neck: Pain causes, osteopathic options. Practical Pain Management. 2020;20(2):54-56.
- See also: Related Info — http://www.pcom.edu